CLINICAL TRIAL: NCT01946243
Title: The Feasibility and Reliability of Utilizing Commercially Available Quantitative Analysis Software as an Adjunct to the Clinical Qualitative Interpretation of Amyvid Brain Scans
Brief Title: The Feasibility of Florbetapir Quantitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-QP01
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physician Readers (Experimental): Physician readers will interpret Amyvid scans using qualitative analysis followed by the use of quantitation. No subjects will be exposed to Florbetapir F 18 as part of this study.
  Interventions: Drug: Florbetapir F18

INTERVENTIONS:
Drug: Florbetapir F18 — No Florbetapir F 18 will be administered in this study.
  Other Names: Amyvid; 18F-AV-45; florbetapir

SUMMARY:
The overall objective of the study is to assess the feasibility of implementing a quantitative process of florbetapir F 18 scan interpretation. The hypothesis is that the use of quantitative analysis will increase the accuracy of florbetapir F 18 scan interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Readers have undergone Amyvid reader training
* Readers have minimal experience with quantitation of amyloid PET scans

Exclusion Criteria:

* Readers have previously been trained to quantitate amyloid PET scans

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals, Inc.
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Florbetapir PET Scans: No subjects were enrolled in this study. Readers interpreted 96 Florbetapir scans from subjects enrolled in previous studies (A07[NCT00857415]/A16[NCT01447719] and A17[NCT01400425]). Scans used in the study included 46 scans with autopsy (A07/A16) and 50 randomly selected non-autopsy scans (A17).
Period: Overall Study
Arm/Group | Florbetapir PET Scans
Started | 96
Completed | 96
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Florbetapir PET Scans
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.9 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Black or African American | 5
  White | 89
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Accuracy (MIMNeuro Software, Low Accuracy Readers)
Description: Evaluate whether the addition of quantitation as an adjunct to qualitative interpretations (VisQ) significantly improved the total accuracy of Amyvid scan interpretation in lower accuracy readers. Only the 46 scans with autopsy from A07/A16 are used for this outcome measure.
Time Frame: Scan acquired 50-60 min post-injection
Measure: Mean (Standard Error); unit: Percent Accuracy
Groups:
- Qualitative: Qualitative scan interpretation only
- VisQ: Quantitation as an adjunct to qualitative scan interpretation
- Change: Change = VisQ - Qualitative
Arm/Group | Qualitative | VisQ | Change
Number analyzed (Participants) | 46 | 46 | 46
Percent Accuracy | 81.7 (2.4) | 88.8 (3.1) | 7.1 (1.5)
Statistical Analysis 1: Comparison: Change; Paired t-test to test whether the change is equal to zero or not; Test type: Superiority or Other; p = 0.0029, t-test, 2 sided

2. Secondary Outcome: Change in Total Accuracy (MIMNeuro Software, All Readers)
Description: Evaluate whether the total accuracy of Amyvid VisQ interpretation was non-inferior to the qualitative scan interpretation alone. Only the 46 scans with autopsy from A07/A16 are used for this outcome measure.
Time Frame: Scan acquired 50-60 min post-injection
Measure: Mean (Standard Error); unit: Percent Accuracy
Arm/Group | Qualitative | VisQ | Change
Number analyzed (Participants) | 46 | 46 | 46
Percent Accuracy | 89.5 (1.4) | 93.8 (1.2) | 4.2 (0.7)
Statistical Analysis 1: Comparison: Change; Test type: Non-Inferiority or Equivalence — Non-inferiority demonstrated if the lower bound of the one-sided 97.5% confidence interval is greater than -3%; Mean Difference (Net) = 4.2, 97.5% CI 1-sided [lower limit 2.7] — Units: Percent Accuracy

3. Secondary Outcome: Change in Reliability (MIMNeuro Software)
Description: Evaluate whether VisQ interpretation significantly improved the reliability of Amyvid scan interpretation compared with qualitative scan interpretation alone. The scan interpretation reliability will be evaluated using Fleiss' Kappa statistics.
Time Frame: Scan acquired 50-60 min post-injection
Measure: Number (95% Confidence Interval); unit: Fleiss Kappa
Arm/Group | Qualitative | VisQ | Change
Number analyzed (Participants) | 96 | 96 | 96
Fleiss Kappa
  All study cases | 0.72 [0.710 to 0.737] | 0.79 [0.774 to 0.801] | 0.06 [0.018 to 0.112]
  Autopsy cases | 0.73 [0.709 to 0.747] | 0.81 [0.787 to 0.825] | 0.08 [0.005 to 0.151]
  Non-autopsy cases | 0.72 [0.700 to 0.737] | 0.77 [0.752 to 0.789] | 0.05 [-0.013 to 0.113]
Statistical Analysis 1: Comparison: Change; Superiority demonstrated if lower bound of two-sided 95% confidence interval (CI) greater than 0, for the change in kappa statistic; Test type: Superiority or Other; lower bound of two-sided 95% CI = 0.06, 95% CI 2-sided [0.018 to 0.112]

4. Secondary Outcome: Change in Total Accuracy (Siemens Syngo.PET Software, Experimental Arm All Readers)
Description: as for outcome 2
Time Frame: Scan acquired 50-60 min post-injection
Measure: Mean (Standard Error); unit: Percent Accuracy
Arm/Group | Qualitative | VisQ | Change
Number analyzed (Participants) | 46 | 46 | 46
Percent Accuracy | 91.6 (0.8) | 93.9 (0.7) | 2.3 (0.7)
Statistical Analysis 1: Comparison: Change; Test type: Non-Inferiority or Equivalence — Non-inferiority demonstrated if the lower bound of the one-sided 97.5% confidence interval is greater than -3%; Mean Difference (Net) = 2.3, 97.5% CI 1-sided [lower limit 0.8] — Units: Percent Accuracy

5. Secondary Outcome: Change in Reliability (Siemens Syngo.PET Software)
Description: Evaluate whether VisQ interpretation significantly improved the reliability of Amyvid scan interpretation compared with qualitative scan interpretations alone. The scan interpretation reliability will be evaluated using Fleiss' Kappa statistics.
Time Frame: Scan acquired 50-60 min post-injection
Measure: Number (95% Confidence Interval); unit: Fleiss Kappa
Arm/Group | Qualitative | VisQ | Change
Number analyzed (Participants) | 96 | 96 | 96
Fleiss Kappa
  All study cases | 0.75 [0.738 to 0.761] | 0.82 [0.805 to 0.827] | 0.07 [0.007 to 0.125]
  Autopsy cases | 0.76 [0.749 to 0.781] | 0.80 [0.785 to 0.817] | 0.04 [-0.046 to 0.112]
  Non-autopsy cases | 0.73 [0.718 to 0.749] | 0.83 [0.815 to 0.846] | 0.10 [0.008 to 0.187]
Statistical Analysis 1: Comparison: Change; Superiority demonstrated if lower bound of two-sided 95% CI greater than 0, for the change in kappa statistic; Test type: Superiority or Other; p = 0.0280, Monte Carlo test; lower bound of two-sided 95% CI = 0.07, 95% CI 2-sided [0.007 to 0.125]

6. Primary Outcome: Change in Total Accuracy (Siemens Syngo.PET Software, Experimental Arm Low Accuracy Readers)
Description: as for outcome 1
Time Frame: Scan acquired 50-60 min post-injection
Measure: Mean (Standard Error); unit: Percent Accuracy
Arm/Group | Qualitative | VisQ | Change
Number analyzed (Participants) | 46 | 46 | 46
Percent Accuracy | 87.0 (1.0) | 91.8 (1.1) | 4.9 (1.1)
Statistical Analysis 1: Comparison: Change; Paired t-test to test whether the change is equal to zero or not; Test type: Superiority or Other; p = 0.0025, t-test, 2 sided

ADVERSE EVENTS:
Description: No subjects received florbetapir in this study. This study consisted of re-reads of scans previously acquired in other clinical studies (A07, A16, and A17).
Groups:
- Florbetapir PET Scans: No subjects received florbetapir in this study. This study consisted of re-reads of scans previously acquired in other clinical studies (A07/A16 and A17).
Arm/Group | Florbetapir PET Scans
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No conclusions can be drawn regarding the relative performance of software packages (different readers) or on impact of additional qualitative practice on quantitative interpretation results (Vis Q always after Qualitative).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes